CLINICAL TRIAL: NCT03761758
Title: Tolerability of a Novel Spectacle Design With Reduced Peripheral Contrast
Acronym: WALNUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: P/639/18/SG
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Lens Design 1 (Experimental): Spectacle lenses design 1, fitted into spectacle frames
  Interventions: Device: Spectacle lenses
- Lens Design 2 (Experimental): Spectacle lenses design 2, fitted into spectacle frames
  Interventions: Device: Spectacle lenses
- Lens Design 3 (Experimental): Spectacle lenses design 3, fitted into spectacle frames
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Spectacle lenses — Spectacle lenses with clear central apertures

SUMMARY:
Prospective, randomized, subject-masked 3-arm clinical study to assess the pediatric acceptability across three iterations of a novel spectacle lens design.

DETAILED DESCRIPTION:
This feasibility study was conducted to assess the performance of three experimental spectacle lens designs (spectacle lenses) in children between 6 and 9 years of age with myopia.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 6 and 12 years
* Myopia between -1.00 and -4.00 D

Exclusion Criteria:

* Participating in any clinical or other research study
* Contact lens wearer

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Distance Visual Acuity | 2 weeks
  Measurement of best corrected distance visual acuity
Contrast Sensitivity | 2 weeks
  Measurement of contrast sensitivity
Subjective Responses | 2 weeks
  Assessment of subject responses related to wear time of spectacles

CONTACTS AND LOCATIONS:
Overall Officials: Joe Rappon, OD, MS, Study Director — SightGlass Vision
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No